CLINICAL TRIAL: NCT05137730
Title: A Randomized, Open-label, Single-center, Single-dose Study to Evaluate the Relative Bioavailability of a New Formulation Compared With the Approved Formulation of Recombinant Human Parathyroid Hormone (rhPTH[1-84]) and to Assess Dose Linearity of the New Formulation in Healthy Subjects
Brief Title: A Study of Relative Bioavailability of a New Formulation Compared With the Approved Formulation of rhPTH [1-84] and to Find Out Dose Linearity of the New Formulation in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-834-1001
Record Dates: First submitted 2021-11-25; First posted 2021-11-30 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part I: Sequence AB (Experimental): Participants will receive a single SC injection of 100 microgram (mcg) rhPTH(1-84) (Formulation A) on Day 1 of treatment period 1 followed by 100 mcg rhPTH(1-84) (Formulation B) on Day 1 of treatment period 2. A washout period of 96 hours will be maintained between each treatment period.
  Interventions: Drug: rhPTH(1-84)
- Part I: Sequence BA (Experimental): Participants will receive a single SC injection of 100 microgram (mcg) rhPTH(1-84) (Formulation B) on Day 1 of treatment period 1 followed by 100 mcg rhPTH(1-84) (Formulation A) on Day 1 of treatment period 2. A washout period of 96 hours will be maintained between each treatment period.
  Interventions: Drug: rhPTH(1-84)
- Part II: Sequence CDEF (Experimental): Participants will receive a single SC injection of 25 mcg (dose C) rhPTH(1-84) on Day 1 of treatment period 1 followed by 50 mcg (dose D) rhPTH(1-84) on Day 1 of treatment period 2 followed by 75 mcg (dose E) rhPTH(1-84) on Day 1 of treatment period 3 followed 200 mcg (dose F) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours will be maintained between each treatment period 1,2,3 and 4.
  Interventions: Drug: rhPTH(1-84)
- Part II: Sequence DFCE (Experimental): Participants will receive a single SC injection of 50 mcg (dose D) rhPTH(1-84) on Day 1 of treatment period 1 followed by 200 mcg (dose F) rhPTH(1-84) on Day 1 of treatment period 2 followed by 25 mcg (dose C) rhPTH(1-84) on Day 1 of treatment period 3 followed by 75 mcg (dose E) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours will be maintained between each treatment period 1,2,3 and 4.
  Interventions: Drug: rhPTH(1-84)
- Part II: Sequence ECFD (Experimental): Participants will receive a single SC injection of 75 mcg (dose E) rhPTH(1-84) on Day 1 of treatment period 1 followed by 25 mcg (dose C) rhPTH(1-84) on Day 1 of treatment period 2 followed by 200 mcg (dose F) rhPTH(1-84) on Day 1 of treatment period 3 followed by 50 mcg (dose D) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours will be maintained between each treatment period 1,2,3 and 4.
  Interventions: Drug: rhPTH(1-84)
- Part II: Sequence FEDC (Experimental): Participants will receive a single SC injection of 200 mcg (dose F) rhPTH(1-84) on Day 1 of treatment period 1 followed by 75 mcg (dose E) rhPTH(1-84) on Day 1 of treatment period 2 followed by 50 mcg (dose D) rhPTH(1-84) on Day 1 of treatment period 3 followed by 25 mcg (dose C) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours will be maintained between each treatment period 1,2,3 and 4.
  Interventions: Drug: rhPTH(1-84)

INTERVENTIONS:
Drug: rhPTH(1-84) — Participants in both part I and part II of the study will receive a single SC injection of rhPTH(1-84) depending upon the treatment sequence allocation on Day 1 of each treatment period.
  Other Names: Recombinant Human Parathyroid Hormone

SUMMARY:
The main aim of Part I of this study is to evaluate the relative bioavailability of a new formulation compared with the approved formulation when a single dose of rhPTH(1-84) is given to healthy volunteers. Bioavailability is the ability of a drug to be absorbed and used by the body. In Part II, the main aim is to assess the dose linearity of the new formulation.

Participants will receive 2 doses in Part I and 4 doses in Part II.

Participants need to visit their doctor approximately 14 days and 30 days after the last dose of study drug.

DETAILED DESCRIPTION:
This study will be conducted in two parts (Part I and Part II). Part I consists of two treatment periods with 2 sequences and part II consists of four treatment periods with 4 sequences. In Part I, relative bioavailability of Formulation A (Test: 100 microgram [mcg] rhPTH[1-84]) will be compared with Formulation B (Reference: 100 mcg rhPTH[1-84]). In Part II, dose linearity of the new formulation, Formulation A, of rhPTH (1-84) will be assessed based on 4 different dose levels as dose c - f (dose c = 25 mcg, dose d = 50 mcg, dose e = 75 mcg and f = 200 mcg). Both parts may be conducted concurrently.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill all of the following inclusion criteria to be eligible for participation in the study:

* Healthy, adult, male or female, 18-65 years of age, inclusive, at screening. Attempts will be made to enroll at least 20% of each sex in each study part.
* Continuous non-smoker who has not used nicotine containing products for at least 90 days prior to the first dosing and throughout the study, based on participant self-reporting.
* Body mass index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m2) at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the Investigator or designee including the following:

  * Serum calcium, parathyroid hormone (PTH), phosphate, and magnesium within laboratory normal limits at screening and check-in.
  * Vitamin D (1,25(OH)2D3) levels between lower limit of normal and up to 1.5x Upper Limit of Normal (ULN).
  * Seated blood pressure Beats per minute (bpm) is >= 89/49 millimeters of mercury (mmHg) and <=139/89 mmHg at screening.
  * Seated pulse rate is >=40 bpm and <=99 bpm at screening.
  * QTcF interval is <=450 millisecond (msec) (males) or <= 470 msec (females) or ECG findings considered normal or not clinically significant by the Investigator or designee at screening.
  * Estimated creatinine clearance >= 80 milliliter per minute (mL/minute) at screening.
* Agrees to comply with any applicable contraceptive requirements of the protocol.
* Understands the study procedures in the ICF, be able to voluntarily provide written, signed, and dated informed consent, and be willing and able to comply with the protocol.

Exclusion Criteria:

Participants must not be enrolled in the study if they meet any of the following criteria:

* Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study in the opinion of the Investigator or designee.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the study drug, or clinical or laboratory assessments.
* Participants who are at increased baseline risk for osteosarcoma such as participants with Paget's disease of bone or unexplained elevations of alkaline phosphatase (ALP), hereditary disorders predisposing to osteosarcoma or a prior history of external beam or implant radiation therapy involving the skeleton.
* History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History or presence of alcoholism or drug abuse, in the opinion of the Investigator or designee, within the past 2 years prior to the first dosing.
* Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day. (1 alcohol unit=1 beer or 1 wine (5 ounces (oz)/150 in milliliters (mL) or 1 liquor (1.5 oz/40 mL) or 0.75 oz alcohol).
* Positive urine drug or alcohol results at screening or check-in.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
* History of abnormalities of calcium homeostasis including hyperparathyroidism, hypoparathyroidism, hyperthyroidism, Cushing's syndrome, hypercalcemia, hypocalcemia, osteoporosis, or any other calcium disorder.
* Female participants who have a positive pregnancy test or who are lactating.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* Has tattoo(s) or scarring at or near the site of injection or any other condition which may interfere with injection site examination, in the opinion of the Investigator or designee.
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine withdrawal headaches. A unit of caffeine is contained in the following items: one 6 oz (180 mL) cup of coffee, two 12 oz (360 mL) cans of cola, one 12 oz cup of tea, three 1 oz (85 g) chocolate bars.
* Prior screen failure, randomization, participation, or enrollment in this study or prior exposure to any exogenous PTH, PTH fragments or analogs 3 months prior to dosing with rhPTH(1-84).
* Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements) Medication, Supplements, and Dietary Products) for the prohibited time period.
* Has been on a diet incompatible with the study diet or had any substantial changes in eating habits, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
* Donation of blood or significant blood loss within 60 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.
* Participation in another clinical study within 30 days or 5 half-lives of the study drug prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Treatment Period 1 of the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61aa7cbcf571d4002a64b451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single site in the United States of America from 29 November 2021 (first participant first visit) and 15 April 2022 (last participant last visit).
Pre-assignment Details: Study was conducted in 2 parts: Part 1 (To Assess Relative Bioavailability) and Part 2 (Dose Linearity). A total of 96 participants (84 participants in Part I and 12 participants in Part II) were enrolled in this study.
Groups:
- Part I: Sequence AB: Participants received a single subcutaneous (SC) injection of 100 microgram (mcg) rhPTH(1-84) (Treatment A) on Day 1 of treatment period 1 followed by 100 mcg rhPTH (1-84) (Treatment B) on Day 1 of treatment period 2. A washout period of 96 hours was maintained between treatment periods 1 and 2.
- Part I: Sequence BA: Participants received a single SC injection of 100 mcg rhPTH(1-84) (Treatment B) on Day 1 of treatment period 1 followed by 100 mcg rhPTH(1-84) (Treatment A) on Day 1 of treatment period 2. A washout period of 96 hours was maintained between treatment periods 1 and 2.
- Part II: Sequence CDEF: Participants received a single SC injection of 25 mcg (Treatment C) rhPTH(1-84) on Day 1 of treatment period 1 followed by 50 mcg (Treatment D) rhPTH(1-84) on Day 1 of treatment period 2 followed by 75 mcg (Treatment E) rhPTH(1-84) on Day 1 of treatment period 3 followed by 200 mcg (Treatment F) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours was maintained between each treatment periods 1, 2, 3 and 4.
- Part II: Sequence DFCE: Participants received a single SC injection of 50 mcg (Treatment D) rhPTH(1-84) on Day 1 of treatment period 1 followed by 200 mcg (Treatment F) rhPTH(1-84) on Day 1 of treatment period 2 followed by 25 mcg (Treatment C) rhPTH(1-84) on Day 1 of treatment period 3 followed by 75 mcg (Treatment E) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours was maintained between each treatment periods 1, 2, 3 and 4.
- Part II: Sequence ECFD: Participants received a single SC injection of 75 mcg rhPTH(1-84) (Treatment E) on Day 1 of treatment period 1 followed by 25 mcg rhPTH(1-84) (Treatment C) on Day 1 of treatment period 2 followed by 200 mcg rhPTH(1-84) (Treatment F) on Day 1 of treatment period 3 followed by 50 mcg rhPTH(1-84) (Treatment D) on Day 1 of treatment period 4. A washout period of 48 hours was maintained between each treatment periods 1, 2, 3 and 4.
- Part II: Sequence FEDC: Participants received a single SC injection of 200 mcg (Treatment F) rhPTH(1-84) on Day 1 of treatment period 1 followed by 75 mcg (Treatment E) rhPTH(1-84) on Day 1 of treatment period 2 followed by 50 mcg (Treatment D) rhPTH(1-84) on Day 1 of treatment period 3 followed by 25 mcg (Treatment C) rhPTH(1-84) on Day 1 of treatment period 4. A washout period of 48 hours was maintained between each treatment periods 1, 2, 3 and 4.
Period: Part I: Treatment Period 1 (1 Day)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 42 | 42 | 0 | 0 | 0 | 0
Completed | 42 | 42 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I: Washout Period 1 (96 Hours)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 42 | 42 | 0 | 0 | 0 | 0
Completed | 42 | 42 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I: Treatment Period 2 (1 Day)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 42 | 42 | 0 | 0 | 0 | 0
Completed | 42 | 42 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Treatment Period 1 (1 Day)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Washout Period 1 (48 Hours)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Treatment Period 2 (1 Day)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Washout Period 2 (48 Hours)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Treatment Period 3 (1 Day)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Washout Period 3 (48 Hours)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II: Treatment Period 4 (1 Day)
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC
Started | 0 | 0 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least one dose of the study drug.
Groups:
- Part I: Sequence AB: Participants received a single SC injection of 100 mcg rhPTH(1-84) (Treatment A) on Day 1 of treatment period 1 followed by 100 mcg rhPTH (1-84) (Treatment B) on Day 1 of treatment period 2. A washout period of 96 hours was maintained between treatment periods 1 and 2.
- Total: Total of all reporting groups
Arm/Group | Part I: Sequence AB | Part I: Sequence BA | Part II: Sequence CDEF | Part II: Sequence DFCE | Part II: Sequence ECFD | Part II: Sequence FEDC | Total
Number analyzed (Participants) | 42 | 42 | 3 | 3 | 3 | 3 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.37) | 45.3 (12.24) | 36.7 (8.14) | 38.0 (4.36) | 45.7 (5.51) | 40.0 (6.24) | 43.0 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 1 | 1 | 2 | 1 | 56
  Male | 15 | 18 | 2 | 2 | 1 | 2 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 30 | 3 | 2 | 2 | 2 | 74
  Not Hispanic or Latino | 7 | 12 | 0 | 1 | 1 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 0 | 0 | 1 | 5
  White | 37 | 36 | 3 | 3 | 3 | 1 | 83
  More than one race | 1 | 3 | 0 | 0 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part I: Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of rhPTH (1-84)
Description: AUClast was a measure of the total amount of drug in the plasma from time zero to time of the last measurable concentration.
Time Frame: Pre-dose, 0.08, 0.16, 0.33, 0.5, 0.75, 1.0, 1.25,1.5,2.0, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours post dose
Population: Pharmacokinetic (PK) Set included all participants who had at least one measurable predose (baseline) and one postdose concentration of parathyroid hormone (PTH). Data was collected and analyzed as per individual treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter (pg*hr/ml)
Groups:
- Part I: Treatment A: Participants received a single SC injection of 100 mcg rhPTH(1-84) (Treatment A) on Day 1 of one of the two treatment periods.
- Part I: Treatment B: Participants received a single SC injection of 100 mcg rhPTH(1-84) (Treatment B) on Day 1 of one of the two treatment periods.
Arm/Group | Part I: Treatment A | Part I: Treatment B
Number analyzed (Participants) | 84 | 84
picogram*hour/milliliter (pg*hr/ml) | 471.9 (57.4) | 603.1 (50.3)
Statistical Analysis 1: Comparison: Part I: Treatment A vs Part I: Treatment B; Test type: Other; Ratio of geometric least squares means = 0.78, 90% CI 2-sided [0.7109 to 0.8611] — Least squares means (LSMs) were calculated by exponentiating the LSMs derived from the linear mixed effects model

2. Primary Outcome: Part II: Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of rhPTH (1-84)
Description: as for outcome 1
Time Frame: Pre-dose, 0.08, 0.16, 0.33, 0.5, 0.75, 1.0, 1.25,1.5,2.0, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours post dose
Population: Pharmacokinetic (PK) Set included all participants who had at least one measurable predose (baseline) and one postdose concentration of parathyroid hormone (PTH). Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. Data was collected and analyzed as per individual treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/ml
Groups:
- Part II: Treatment C: Participants received a single SC injection of 25 mcg (Treatment C) rhPTH(1-84) on Day 1 of one of the four treatment periods.
- Part II: Treatment D: Participants received a single SC injection of 50 mcg (Treatment D) rhPTH(1-84) on Day 1 of one of the four treatment periods.
- Part II: Treatment E: Participants received a single SC injection of 75 mcg (Treatment E) rhPTH(1-84) on Day 1 of one of the four treatment periods.
- Part II: Treatment F: Participants received a single SC injection of 200 mcg (Treatment F) rhPTH(1-84) on Day 1 of one of the four treatment periods.
Arm/Group | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 11 | 12 | 12 | 12
pg*hr/ml | 44.34 (161.7) | 97.74 (123.4) | 259.2 (57.5) | 1009 (61.3)
Statistical Analysis 1: Comparison: Part II: Treatment C vs Part II: Treatment D vs Part II: Treatment E vs Part II: Treatment F; A linear regression model was used, including sequence and period as fixed effects, subject within sequence as a random effect, and ln(dose) as a covariate; Test type: Other; Dose effect = 1.5395, 95% CI 2-sided [1.2929 to 1.7862], Standard Error of Mean 0.1210

3. Primary Outcome: Part I: Area Under the Plasma Concentration- Time Curve From Time Zero to Infinity (AUCinf) of rhPTH(1-84)
Description: AUCinf was the area under the curve extrapolated to infinity, calculated using the observed value of the last non-zero concentration. AUC was be used as a measure of drug exposure. It was derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Pre-dose, 0.08, 0.16, 0.33, 0.5, 0.75, 1.0, 1.25,1.5,2.0, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours post dose
Population: PK Set included all participants who had at least one measurable predose (baseline) and one postdose concentration of parathyroid hormone (PTH). Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. Data was collected and analyzed as per individual treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/ml
Arm/Group | Part I: Treatment A | Part I: Treatment B
Number analyzed (Participants) | 73 | 79
pg*hr/ml | 559.7 (53.2) | 663.7 (44.0)
Statistical Analysis 1: Comparison: Part I: Treatment A vs Part I: Treatment B; Test type: Other; Ratio of geometric least squares means = 0.84, 90% CI 2-sided [0.7576 to 0.9375] — LSMs were calculated by exponentiating the LSMs derived from the linear mixed effects model

4. Primary Outcome: Part II: Area Under the Plasma Concentration- Time Curve From Time Zero to Infinity (AUCinf) of rhPTH(1-84)
Description: as for outcome 3
Time Frame: Pre-dose, 0.08, 0.16, 0.33, 0.5, 0.75, 1.0, 1.25,1.5,2.0, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours post dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/ml
Arm/Group | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 2 | 6 | 7 | 11
pg*hr/ml | 83.91 (19.5) | 217.0 (33.2) | 364.7 (39.0) | 1117 (59.6)
Statistical Analysis 1: Comparison: Part II: Treatment C vs Part II: Treatment D vs Part II: Treatment E vs Part II: Treatment F; A linear regression model using was used, including sequence and period as fixed effects, subject within sequence as a random effect, and ln(dose) as a covariate; Test type: Other; Dose effect = 1.2823, 95% CI 2-sided [1.0431 to 1.5215], Standard Error of Mean 0.1072

5. Primary Outcome: Part I: Maximum Observed Plasma Concentration (Cmax) of rhPTH(1-84)
Description: Cmax referred to the maximum (or peak) concentration that a drug achieved in the body after the drug had been administrated.
Time Frame: Pre-dose, 0.08, 0.16, 0.33, 0.5, 0.75, 1.0, 1.25,1.5,2.0, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours post dose
Population: PK Set included all participants who had at least one measurable predose (baseline) and one postdose concentration of parathyroid hormone (PTH). Data was collected and analyzed as per individual treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/ml)
Groups:
- Part I: Treatment A: Participants received a single SC injection of 100 mcg rhPTH(1-84) (Treatment A) on Day 1 of one of the four treatment periods.
Arm/Group | Part I: Treatment A | Part I: Treatment B
Number analyzed (Participants) | 84 | 84
picogram per milliliter (pg/ml) | 150.8 (53.2) | 185.1 (52.7)
Statistical Analysis 1: Comparison: Part I: Treatment A vs Part I: Treatment B; Test type: Other; Ratio of geometric least squares means = 0.81, 90% CI 2-sided [0.7462 to 0.8893] — LSMs were calculated by exponentiating the LSMs derived from the linear mixed effects model

6. Primary Outcome: Part II: Maximum Observed Plasma Concentration (Cmax) of rhPTH(1-84)
Description: as for outcome 5
Time Frame: Pre-dose, 0.08, 0.16, 0.33, 0.5, 0.75, 1.0, 1.25,1.5,2.0, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours post dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 11 | 12 | 12 | 12
pg/ml | 28.05 (50.4) | 43.06 (47.5) | 77.46 (55.8) | 250.2 (41.5)
Statistical Analysis 1: Comparison: Part II: Treatment C vs Part II: Treatment D vs Part II: Treatment E vs Part II: Treatment F; [analysis description as in outcome 2, analysis 1]; Test type: Other; Dose effect = 1.0937, 95% CI 2-sided [0.9380 to 1.2493], Standard Error of Mean 0.0763

7. Secondary Outcome: Part I and II: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE was an adverse event with a start date on or after the first dose of Investigational product (IP), or a start date before the date of the first dose of IP but increased in severity on or after the date of the first dose of IP. Number of participants with TEAEs was reported.
Time Frame: From start of study drug administration up to Day 34
Population: Safety set included all participants who received at least one dose of the study drug. Data was collected and analyzed as per individual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Treatment A | Part I: Treatment B | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 84 | 84 | 12 | 12 | 12 | 12
Participants | 19 | 15 | 2 | 4 | 3 | 2

8. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Values
Description: Vital sign assessments included systolic and diastolic blood pressure, pulse rate and body temperature. Any change in vital signs which are deemed clinically significant by the investigator were reported.
Time Frame: From start of study drug administration up to Day 34
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Treatment A | Part I: Treatment B | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 84 | 84 | 12 | 12 | 12 | 12
Participants | 1 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part I and II: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters Reported as TEAEs
Description: Any change in ECG assessments which were deemed clinically significant by the investigator were reported.
Time Frame: From start of study drug administration up to Day 34
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Treatment A | Part I: Treatment B | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 84 | 84 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Part I and II: Number of Participants With Clinically Significant Changes in Clinical Laboratory Values
Description: Clinical laboratory tests included hematology, chemistry, and urinalysis. Any changes in clinical laboratory results which are deemed clinically significant by the investigator were reported.
Time Frame: From start of study drug administration up to Day 34
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Treatment A | Part I: Treatment B | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
Number analyzed (Participants) | 84 | 84 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 34
Description: Safety set included all participants who received at least one dose of the study drug.
Arm/Group | Part I: Treatment A | Part I: Treatment B | Part II: Treatment C | Part II: Treatment D | Part II: Treatment E | Part II: Treatment F
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/84 | 9/84 | 2/12 | 4/12 | 3/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Treatment A (N=84) | Part I: Treatment B (N=84) | Part II: Treatment C (N=12) | Part II: Treatment D (N=12) | Part II: Treatment E (N=12) | Part II: Treatment F (N=12)
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 7 | 4 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT05137730/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT05137730/SAP_001.pdf